CLINICAL TRIAL: NCT01087528
Title: Evaluation of PillCam™ Colon 2 in Visualization of the Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MA-202
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2012-06-08 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Colonic Diseases; Bowel Diseases
Keywords: Colonic Diseases; bowel diseases; large bowel diseases
MeSH Terms: conditions — Colonic Diseases; Intestinal Diseases | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Subjects that are indicated for colonoscopy, who are suspected or known to suffer from large bowel diseases.
  Interventions: Device: PillCam™ (Capsule Endoscopy) Colon 2 capsule

INTERVENTIONS:
Device: PillCam™ (Capsule Endoscopy) Colon 2 capsule — Medical Device

SUMMARY:
To evaluate the performance of PillCam COLON 2 in regards to detection of patients with polyps where colonoscopy is considered as the gold standard reference.

DETAILED DESCRIPTION:
Standard evaluation of subjects with suspected colon diseases includes endoscopic imaging by colonoscopy and radiology testing such as: air-contrast barium enema, abdominal/pelvic CT, or virtual colonoscopy.

The Given® Diagnostic System offers an alternative approach for endoscopic visualization of the colon. Advantages of the Given® Diagnostic System include the elimination of the need for conscious sedation, the minimally invasive, painless nature of the exam, and the ability to pursue normal daily activities immediately following the procedure . Furthermore, compared to standard colonoscopy, the Given® Diagnostic System may be more readily accepted by the subjects, thereby improving subjects' willingness to undergo a diagnostic evaluation of the colon and comply with colorectal cancer screening recommendations.

The PillCam™ SB capsule (formerly M2A® Capsule) that was cleared by the FDA- in August 2001 for small bowel evaluation has been ingested to date by more than 1,000,000 people worldwide and is well accepted by patients and physicians as well as the professional societies. However, adequate visualization of the colon cannot be achieved with the standard PillCam™ SB capsule because of the anatomical and physiological properties of the colon which are significantly different than the small bowel. Moreover, other issues that limit the evaluation of the colonic mucosa by the standard PillCam™ SB procedure include an unsatisfactory level of colon cleanliness and slow progression of the PillCam™ SB capsule through the colon during the desired examination time. Therefore, the development and introduction of a specially designed, customized colon capsule combined with a dedicated capsule colonoscopy procedure protocol will allow for more efficient evaluation of the colonic mucosa. This is expected to improve the capability of the Given® Diagnostic System to detect colonic pathologies and to serve as a diagnostic and screening tool for colonic disease. To date, several clinical studies have been conducted with Given® Diagnostic System and the PillCam™ Colon 1 capsule A pilot multicenter study is currently being conducted with a new Given® Diagnostic System and an advanced generation of the the PillCam™ Colon capsule - PillCam™ Colon 2. Capsule. The new development of Given® Diagnostic System and PillCam™ Colon 2 capsule is primarily aimed to increase sensitivity and specificity for polyp detection.

Further details of the Given® Diagnostic System and PillCam™ Colon 2 capsule can be found in the device description section.

This study is designed to evaluate the performance of the new version of Given® Diagnostic System and PillCam™ Colon 2 capsule in detecting patients with polyps and other colonic lesions as compared to conventional colonoscopy.

ELIGIBILITY:
Inclusion criteria:

* Subject is between the ages of 18-70
* Subject was referred to colonoscopy for at least one of the following reasons:

  * Colorectal cancer screening for age ≥60
  * Clinical symptoms such as: rectal bleeding, hematochezia, melena, positive FOBT, recent change of bowel habits for age ≥50
  * Positive findings in the colon (e.g. Polyp ≥10mm)
  * Personal history of significant polyps( ≥6mm )that were removed at least 3 years ago (3 years and above)

Exclusion criteria

* Age > 70 years
* Subject has dysphagia or any swallowing disorder
* Subject has congestive heart failure
* Subject has known renal disease
* Subject is not eligible for colon preparation due to the presence of underlying conditions based on the clinical judgment of the investigator
* Subject has any allergy or other known contraindication to the medications used in the study
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
* Subject has a cardiac pacemaker or other implanted electro medical device.
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject with any condition believed to have an increased risk for capsule retention such as Crohn's disease, intestinal tumors, radiation enteritis, incomplete colonoscopies due to obstructions or NSAID enteropathy,
* Subject with gastrointestinal motility disorders
* Subject has known delayed gastric emptying
* Subject has any condition, which precludes compliance with study and/or device instructions.
* Women who are either pregnant at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
* Subject suffers from life threatening conditions
* Subject currently participating in another clinical study
* Age>70

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Rex, Dr., Principal Investigator — Division of Gastroenterology, Indiana University Medical Center
Locations (4):
- United States (4):
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of North Carolina, Chapel Hill, North Carolina
  - Digestive Care, Inc., Beavercreek, Ohio
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia

REFERENCES:
- [Derived] Morgan DR, Malik PR, Romeo DP, Rex DK. Initial US evaluation of second-generation capsule colonoscopy for detecting colon polyps. BMJ Open Gastroenterol. 2016 May 3;3(1):e000089. doi: 10.1136/bmjgast-2016-000089. eCollection 2016. PMID 27195129

RESULTS

PARTICIPANT FLOW:
Groups:
- Colon Capsule Endoscopy, Then Standard Colonoscopy: Capsule endoscopy was ingested following colon preparation without colon insufflation or sedation.The purpose was to detect patients with polyps equal or larger than 6mm. Patients subsequently had standard colonoscopy as "gold standard" comparison..
Period: Overall Study
Arm/Group | Colon Capsule Endoscopy, Then Standard Colonoscopy
Started | 51
Completed | 44 (withdrawn from the study prior to any procedure)
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Incomplete CE procedure | 6

BASELINE CHARACTERISTICS:
Arm/Group | Colon Capsule Endoscopy, Then Standard Colonoscopy
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.22 (6.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Detection in Patients With Colonic Polyps - Sensitivity
Description: The accuracy parameters (i.e. sensitivity) were evaluated for detection of patients with polyps equal or larger than 6 mm and for detection of patients with polyps equal or larger than 10 mm by constructing 2X2 matrix (i.e. PCCE-2 performance versus the standard colonoscopy), where sensitivity and specificity, are presented with 95% Cl based on the binomial distribution. Standard colonoscopy is considered the gold standard.
Time Frame: within 7 days
Population: Patients were included in the study due to a referral for colonoscopy for a variety of reasons such as recent change of bowel habits, prior positive findings, rectal bleeding, abdominal pain or a positive FOBT.
Measure: Number (95% Confidence Interval); unit: percentage of sensiivity
Groups:
- PillCam COLON: Ingestible capsule equipped with an endoscope with two imagers, given after bowel preparation and before standard colonoscopy.
Arm/Group | PillCam COLON
Number analyzed (Participants) | 44
percentage of sensiivity
  Patients with Polyp>= 6 mm | 89 [61 to 98]
  Patients with Polyp, >= 10 mm | 100 [46 to 100]

2. Primary Outcome: Accuracy of Detection in Patients With Colonic Polyps - Specificity
Description: The accuracy parameters (i.e. specificity) were evaluated for detection of patients with polyps equal or larger than 6 mm and for detection of patients with polyps equal or larger than 10 mm by constructing 2X2 matrix (i.e. PCCE-2 performance versus the standard colonoscopy), where sensitivity and specificity, are presented with 95% Cl based on the binomial distribution. Standard colonoscopy is considered the gold standard.
Time Frame: within 7 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of specificity
Arm/Group | PillCam COLON
Number analyzed (Participants) | 44
percentage of specificity
  Patients with Polyp>= 6 mm | 43 [36 to 45]
  Patients with Polyp, >= 10 mm | 66 [62 to 66]

3. Secondary Outcome: Diagnostic Yield of PillCam™ COLON 2 in Detecting Colonic Lesions
Description: The diagnostic yield (%) of PCCE-2 and colonoscopy in visualizing a variety of colonic lesion excluding polyps (e.g. inflammation, diverticulosis and bleeding lesions) is provided.
Time Frame: within 7 days
Population: as for outcome 1
Measure: Number; unit: percentage of yield
Groups:
- PillCam COLON; Standard Colonoscopy: All subjects received ingestible capsule equipped with an endoscope with two imagers, given after bowel preparation and before standard colonoscopy. Results compare capsule vs. colonoscopy.
Arm/Group | PillCam COLON | Standard Colonoscopy
Number analyzed (Participants) | 44 | 44
percentage of yield
  %Patients Yield Diverticulosis | 83 | 61
  %Patients Yield Inflamatory | 4.5 | 9
  %Patients Yield Angiodysplasia | 4.5 | 0

4. Secondary Outcome: Percent of Participants With Scoring Index 3 or 4 (Good or Excellent)
Description: Overall colon cleanliness was judged for capsule endoscopy and colonoscopy on a four-point grading index scale as follows:
  1. poor cleansing level (Large amount of fecal residue.)
  2. fair cleansing level (Enough feces or dark fluid present to preclude a completely reliable examination.)
  3. good cleansing level (Small amount of feces or dark fluid, but not enough to interfere with examination.)
  4. excellent cleansing level (No more than small bits of adherent feces.)
Time Frame: within 7 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PillCam COLON | Standard Colonoscopy
Number analyzed (Participants) | 44 | 44
percentage of participants
  Overall | 61 [46 to 75] | 86 [73 to 94]
  Rectum | 43 [31 to 67] | 92 [81 to 98]
  Decending Colon | 83 [67 to 93] | 86 [73 to 94]
  Transverse Colon | 59 [42 to 74] | 82 [69 to 91]
  Ascending Colon | 61 [46 to 75] | 88 [75 to 95]
  Cecum | 63 [47 to 76] | 88 [75 to 95]

5. Secondary Outcome: Capsule Excretion Time
Description: Capsule excretion time is defined as the duration of ingestion to capsule excretion time. The distribution of excretion times were categorized as follows:
  * capsule excreted within 4 hours
  * capsule excreted within 6 hours
  * capsule excreted within 8 hours
  * capsule excreted 8 hours and above
Time Frame: within 7 days
Population: All subject who ingested the capsule were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | PillCam COLON
Number analyzed (Participants) | 50
Participants
  excreated <4hr | 8
  excreated >4h and <6hr | 13
  excreated >6hr ans <8hr | 8
  excreted 8hr+ | 21

ADVERSE EVENTS:
Arm/Group | Colon Capsule Endoscopy, Then Standard Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 3/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colon Capsule Endoscopy, Then Standard Colonoscopy (N=51)
bruising to abdomen (Gastrointestinal disorders) | 1 (1)
Left eye pain (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No